CLINICAL TRIAL: NCT05249452
Title: Adding Azathioprine/Hydroxyurea Preconditioning to Alemtuzumab/TBI to Reduce Risk of Graft Failure in Matched Sibling Donor Allogeneic HSCT in Adult Sickle Cell Patients
Brief Title: Adding Azathioprine/Hydroxyurea Preconditioning to Alemtuzumab/TBI to Reduce Risk of Graft Failure in MSD HSCT in Adult SCD Patients
Status: Completed | Type: Observational
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, Erfan Nur, Principal Investigator, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Other Study IDs: W21_160
Record Dates: First submitted 2022-01-06; First posted 2022-02-21 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Sickle Cell Disease
Keywords: Sickle Cell Disease; Allogeneic stem cell transplantation; Mixed chimerism
MeSH Terms: conditions — Anemia, Sickle Cell | interventions — Hydroxyurea

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adult transplant-eligible SCD patients with a MSD: Sickle cell disease patients aged 16 years and older with an available matched sibling donor.
  Interventions: Other: Preconditioning with azathiprine and hydroxyurea (3 months)

INTERVENTIONS:
Other: Preconditioning with azathiprine and hydroxyurea (3 months) — Preconditioning with azathiprine and hydroxyurea (3 months) before alemtuzumab/TBI conditioning and matched sibling donor allogeneic stem cell transplantation.

SUMMARY:
In this study the investigators will prospectively investigate whether the addition of a 3-months long preconditioning with azathioprine to the alemtuzumab/TBI non-myeloablative conditioning results in improved disease-free survival and donor chimerism after allo-SCT in SCD patients. Furthermore, the investigators will evaluate whether azathioprine/hydroxyurea preconditioning leads to more patients being able to taper and discontinue sirolimus at 12 months post-transplantation.

DETAILED DESCRIPTION:
Matched sibling donor (MSD) transplantation with non-myeloablative conditioning (1 mg/kg alemtuzumab and 300 cGy total body irradiation (TBI)) using peripheral blood derived stem cells has shown promising results in adult SCD patients. However, a large part of these patients did not reach complete donor chimerism (especially relatively low T-cell chimerism) with graft failure rates of approximately 13%. Furthermore a significant proportion of sickle cell patients need to continuously use the immunosuppressive medication sirolimus to prevent graft failure due to poor donor T-cell chimerism. Graft failure is more common in sickle cell patients than in patients who are transplanted for hematological malignancies. Due to the continuously active erythropoiesis, patients with hemoglobinopathies, such as thalassemia and SCD, have expanded bone marrow, which negatively affects engraftment. Another reason for graft failure in these patients is a continuously triggered immune system due to chronic hemolysis and inflammation in hemoglobinopathies. To improve engraftment and donor chimerism, a preconditioning with azathioprine (immunosuppressive) and hydroxyurea (suppressing bone marrow expansion) during three months has been added to the actual conditioning with alemtuzumab/TBI. Azathioprine/hydroxyurea preconditioning has been proven effective in allo-SCT in thalassemia.

In this study the investigators will prospectively investigate whether the addition of a 3-months long preconditioning with azathioprine to the alemtuzumab/TBI non-myeloablative conditioning results in improved disease-free survival and donor chimerism after allo-SCT in SCD patients. A secondary objective is to evaluate whether azathioprine/hydroxyurea preconditioning leads to more patients being able to taper and discontinue sirolimus at 12 months post-transplantation.

Protocol was amended: in the case of impending graft rejection, defined as declining T-cell chimerism in combination with new onset cytopenias, a second course of alemtuzumab 1mg/kg can be administered in order to avert overt graft failure.

ELIGIBILITY:
Inclusion Criteria:

* SCD patients with an HLA-identical matched sibling donor eligible for allogeneic stem cell transplantation.
* Age 16 - 60 years
* Good performance status (ECOG 0 or 1; Karnofsky and Lansky 70-100)
* Patients and donors (MSD) must be able to sign consent forms for receiving and donating hematopoietic stem cells respectively. The sibling donor should be willing to donate.
* Patients must be geographically accessible and willing to participate in all stages of treatment.
* Eligible diagnoses: Patients with sickle cell disease such as sickle cell anemia (Hb SS), Hb/Sβ0-thalassemia, Hb/Sβ+-thalassemia, HbSC disease, HbSE disease, HbSD disease and Hemoglobin SO- Arab disease.

Exclusion Criteria:

* Poor performance status (ECOG>1).
* Poor cardiac function: left ventricular ejection fraction<35%.
* Poor pulmonary function: FEV1 and FVC<40% predicted.
* Poor liver function: direct bilirubin >3.1 mg/dl
* HIV-positive
* Women of childbearing potential who currently are pregnant (Beta-HCG+) or who are not practicing adequate contraception.
* Patients who have any debilitating medical or psychiatric illness that would preclude their giving informed consent or their receiving optimal treatment and follow-up. However, patients with history of stroke and significant cognitive deficit, that would preclude giving informed consent or assent will not be excluded, if they have a family member or significant other with Power of Attorney to also consent of their behalf.

Ages: 16 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Sickle cell disease patients, 16 years and older, with an available matched sibling donor.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2018-03-08 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
Disease-free survival | 1 year post-transplantation

SECONDARY OUTCOMES:
Transplantation-related complications | Day 100 post-transplantation
Transplantation-related complications | 1 year post-transplantation
Attenuation of SCD-related organ complications | 1 year post-transplantation
Percentage of donor myeloid chimerism | 2 years post-transplantation
  Using genetic profiles of both the patient and the donor, percentages of myeloid (isolated granulocytes) chimerism will be measured periodically to evaluate the level of engraftment.
Percentage of donor T-cell chimerism | 2 years post-transplantation
  Using genetic profiles of both the patient and the donor, percentages of T-cell (CD3 cells) chimerism will be measured periodically to evaluate the level of engraftment.
Primary graft failure | day 42 post-transplantation
  Defined as never achieving >5% donor whole blood or myeloid chimerism (myeloid is preferable) assessed by bone marrow or peripheral blood chimerism assays by day +42 post-transplant. Second infusion of stem cells is also considered indicative of primary graft failure by day +42 post-transplant.
Secondary graft failure | 2-years post-transplantation
  Defined as < 5% donor whole blood or myeloid chimerism (myeloid is preferable) in peripheral blood or bone marrow beyond day +42 post-transplant in patients with prior documentation of hematopoietic recovery with >5% donor cells by day +42 post-transplant. Second infusion of stem cells is also considered indicative of secondary graft failure.

CONTACTS AND LOCATIONS:
Overall Officials: Erfan Nur, MD, PhD, Principal Investigator — Amsterdam UMC
Locations (1):
- Amsterdam Medical Centre, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Dovern E, Aydin M, Hazenberg MD, Tang MW, Suijk EM, Hoogendoorn GM, Van Tuijn CFJ, Kerkhoffs JL, Rutten CE, Zeerleder SS, de la Fuente J, Biemond BJ, Nur E. Azathioprine/hydroxyurea preconditioning prior to nonmyeloablative matched sibling donor hematopoietic stem cell transplantation in adults with sickle cell disease: A prospective observational cohort study. Am J Hematol. 2024 Aug;99(8):1523-1531. doi: 10.1002/ajh.27360. Epub 2024 May 11. PMID 38733340